CLINICAL TRIAL: NCT06991556
Title: A Phase II, Randomized, Open-label, Multi-center Study of JSB462 (Luxdegalutamide) in Combination With Abiraterone in Adult Male Patients With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Brief Title: An Open-label Study of JSB462 (Luxdegalutamide) in Combination With Abiraterone in Adult Male Patients With Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJSB462C12201; 2024-520156-22-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
Keywords: Interventional; clinical trial; open-label; JSB462; luxdegalutamide; efficacy; safety; tolerability; abiraterone; metastatic hormone-sensitive prostate cancer
MeSH Terms: interventions — abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): JSB462 100 mg QD + abiraterone 1000 mg QD
  Interventions: Drug: JSB462; Drug: Abiraterone
- Arm 2 (Experimental): JSB462 300 mg QD + abiraterone 1000 mg QD
  Interventions: Drug: JSB462; Drug: Abiraterone
- Arm 3 (Active Comparator): abiraterone 1000 mg QD or enzalutamide 160 mg QD
  Interventions: Drug: Abiraterone; Drug: Enzalutamide

INTERVENTIONS:
Drug: JSB462 — JSB462 is administered orally, daily and continuously (100 mg or 300 mg QD) until disease progression per PCWG3-modified RECIST 1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.
  Other Names: luxdegalutamide
  Arms: Arm 1; Arm 2
Drug: Abiraterone — Abiraterone 1000 mg is administered orally, daily and continuously until disease progression per PCWG3-modified RECIST 1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.
Drug: Enzalutamide — Enzalutamide 160 mg is administered orally, daily and continuously until disease progression per PCWG3-modified RECIST 1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.
  Arms: Arm 3

SUMMARY:
This Phase II study aims to evaluate efficacy and safety of the combination of JSB462 (also known as luxdegalutamide) at 100 mg and 300 mg once a day (QD) doses + abiraterone compared with an androgen receptor pathway inhibitor (ARPI, abiraterone or enzalutamide) in participants with metastatic Hormone Sensitive Prostate Cancer (mHSPC) and to select the recommended dose of the combination for phase III. Towards that end, the totality of the efficacy, safety, tolerability and PK data from participants randomized in the study will be evaluated

DETAILED DESCRIPTION:
The study for each participant consists of a Screening period (28 days), a treatment period, a post-treatment safety follow-up (30 days) followed by a long-term follow-up period.

During the treatment period:

* JSB462 is administered from randomization, orally, daily and continuously (100 mg or 300 mg QD) until disease progression per PCWG3-modified RECIST 1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.
* Abiraterone 1000 mg or enzalutamide 160 mg are administered from randomization, orally, daily, and continuously until disease progression per PCWG3-modified RECIST 1.1 as assessed by the investigator, the occurrence of unacceptable toxicities, death, participant decision or investigator decision.

During the post-treatment follow up period:

* Safety follow-Up: After discontinuation of study treatment, all participants will be followed for at least 1 safety follow-up visit (30 days [+/- 7 days] after treatment discontinuation). Subsequent lines of therapy may be administered according to investigator's discretion after treatment discontinuation.
* Long-term follow-up: Starts after the Safety follow-up period and lasts until the end of study. Safety, efficacy and survival information may be collected from participants during this period.

ELIGIBILITY:
Key Inclusion Criteria:

* An Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤2
* Histologically confirmed adenocarcinoma of the prostate. Participants with mixed histology (neuroendocrine) are not eligible
* High-volume mHSPC, defined by the presence of ≥1 metastatic visceral non-nodal lesion and/or ≥4 metastatic bone lesions (with at least one lesion outside the vertebral column and/or pelvis) in imaging exams (CT/MRI or bone scan) according to local radiology assessment by the investigator obtained ≤28 days prior to randomization
* Participants must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L). Ongoing ADT (as defined by prior orchiectomy and/or ongoing GnRH analog/antagonist) for ≤90 days is allowed prior to randomization, provided that PSA zero (PSA level <0.2 ng/ml according to local laboratory as assessed by the investigator) is not achieved prior to randomization.

Key Exclusion Criteria:

* Prior exposure to a second generation ARPI (such as enzalutamide/darolutamide/apalutamide and/or abiraterone) for the treatment of advanced/metastatic disease is not allowed. Prior exposure to ARPI, to taxane chemotherapy (up to 6 cycles) or to RLT in the context of (neo)adjuvant treatment for localized prostate cancer is allowed, if the last dose of this treatment was administered >12 months from randomization. Prior use of a first generation ARPI (such as bicalutamide) in the context of ADT initiation with a GnRH analog is allowed, provided the first generation ARPI was administered for ≤14 days and last dose was administered ≥7 days from randomization.
* Participants with biochemical recurrence only or those without evidence of metastatic disease by radiological imaging (CT/MRI or bone scan) are not eligible

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2032-04-19 (Estimated); Study Completion 2035-11-07 (Estimated)

PRIMARY OUTCOMES:
Prostate Specific Antigen 90 (PSA90) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  Prostate Specific Antigen 90 (PSA90) Rate is defined as the proportion of participants who achieve a ≥90% decrease in PSA from baseline at any timepoint, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between.
Incidence rate of adverse events (AEs) | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  The analysis of adverse events will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Number of participants with dose adjustments | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) will be summarized by treatment arm.
Duration of exposure to study treatment | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  The duration of exposure in weeks to study treatment and for each study treatment component (JSB462, abiraterone and enzalutamide) will be summarized for each study treatment component by means of descriptive statistics using the SAS.

SECONDARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 83 months
  Radiographic Progression Free Survival (rPFS) is defined as the time between randomization and the first occurrence of disease progression (per PCWG3-modified RECIST 1.1 as assessed by the investigator) or death due to any cause
Overall Survival (OS) | From date of randomization until date of death from any cause, assessed up to approximately 83 months
  Overall Survival (OS) is defined as the time between randomization and death due to any cause
Incidence rate of adverse events (AEs) | From date of randomization till 30 days safety fup, assessed up to approximately 83 months
  The analysis of adverse events and laboratory abnormalities will include categorization by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Overall Response Rate (ORR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 83 months
  Overall Response Rate (ORR) is defined as the proportion of participants achieving a confirmed complete response (CR) or partial response (PR) per PCWG3-modified RECIST 1.1 as assessed by the investigator
Disease Control Rate (DCR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 83 months
  Disease Control Rate (DCR) is defined as the proportion of participants achieving a CR, PR or stable disease (SD) per PCWG3-modified RECIST 1.1 as assessed by the investigator
Duration of Response (DOR) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to approximately 83 months
  Duration of Response (DOR) is defined as the time between first documented CR/PR and disease progression or death due to any cause per PCWG3-modified RECIST 1.1 as assessed by the investigator
Time to Response (TTR) | From date of randomization until date of first documented Complete Response (CR) or Partial Response (PR), assessed up to approximately 83 months
  Time to response (TTR) is defined as the time from randomization to the date of first documented CR or PR per PCWG3-modified RECIST 1.1 as assessed by the investigator
Time to soft tissue progression (TTSTP) | From date of randomization until date of soft tissue radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 83 months
  Time to soft tissue progression (TTSTP) is defined as the time from randomization to the date of first documented radiographic soft tissue progression per PCWG3-modified RECIST 1.1 as assessed by the investigator
Prostate Specific Antigen 30 (PSA30) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  Prostate Specific Antigen 30 (PSA30) Rate is defined as the proportion of participants who achieve a ≥30% decrease from baseline at any timepoint, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between
Prostate Specific Antigen 50 (PSA50) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  Prostate Specific Antigen 50 (PSA50) Rate is defined as the proportion of participants who achieve a ≥50% decrease from baseline at any timepoint, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between
Prostate Specific Antigen 0 (PSA0) Rate | From date of randomization till 30 days safety fup, assessed up to approximately 75 months
  Prostate Specific Antigen 0 (PSA0) Rate is defined as the proportion of participants who achieve a PSA level <0.2 ng/ml at any timepoint after start of treatment, confirmed by a second PSA measurement ≥3 weeks without any PSA progression in between
Duration of biochemical response (DBR) | From date of date of first PSA50 response until date of PSA progression or death from any cause, assessed up to approximately 83 months
  Duration of biochemical response (DBR) is defined as the time between PSA90 and/or PSA0 and PSA progression (increase ≥25% in PSA and an absolute increase of ≥2 ng/mL from NADIR) or death due to any cause
Time to first symptomatic skeletal event (TTSSE) | From date of randomization till EOT or death, whichever happens first, assessed up to approximately 83 months
  Time to first symptomatic skeletal event (TTSSE) is defined as the date of randomization to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first
Plasma concentrations of JSB462 and plasma concentrations of its metabolite ARV-767 | Day 1 of Cycles 1 and 2: Pre-dose/0h and Post-dose 4h +/- 1h. Day 1 of Cycles 3 to 8: Pre-dose/0h. End of Treatment Visit (EOT): Anytime. 1 cycle = 28 days.
  JSB462 pharmacokinetic (PK) samples will be obtained and evaluated in all participants at all dose levels in JSB462 treatment arms.
Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | From randomization up till 30 day safety Follow-up, assessed up to approximately 83 months
  The PRO-CTCAE is a patient-reported outcomes measurement system developed by the National Cancer Institute as a companion to the CTCAE. It includes items covering participant-reported symptomatic adverse events (AEs) from the CTCAE. Each symptomatic AE concept has up to three items evaluating frequency, severity, or interference, focused on the study population and treatment regimens.
  Participants respond on a 5-point scale for each item:
  * Frequency: Never, Rarely, Occasionally, Frequently, Almost constantly
  * Severity: None, Mild, Moderate, Severe, Very severe
  * Interference: Not at all, A little bit, Somewhat, Quite a bit, Very much
  The past 7-day recall version is used, focusing on relevant symptoms like fatigue, diarrhea, and hot flashes.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (14):
  - University of California San Diego - Moores Cancer Center, La Jolla, California
  - Saint Johns Cancer Institute, Santa Monica, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Emory University School of Medicine-Winship Cancer Institute, Atlanta, Georgia
  - Mass General Hospital, Boston, Massachusetts
  - XCancer Omaha LLC, Omaha, Nebraska
  - Perlmutter Cancer Centre, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Urology San Antonio, San Antonio, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutch Cancer Research, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Beijing, Chaoyang
  - Novartis Investigative Site, Beijing
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (4):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Quint-Fonsegrives
  - Novartis Investigative Site, Suresnes
- Germany (3):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Nürtingen
- Italy (3):
  - Novartis Investigative Site, Asti, AT
  - Novartis Investigative Site, Trento, TN
  - Novartis Investigative Site, Verona, VR
- Netherlands (4):
  - Novartis Investigative Site, Zwolle, Overijssel
  - Novartis Investigative Site, Dordrecht, South Holland
  - Novartis Investigative Site, Hoofddorp
  - Novartis Investigative Site, Schiedam
- Poland (4):
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Oświęcim
  - Novartis Investigative Site, Skorzewo
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com